CLINICAL TRIAL: NCT04242706
Title: VITAL - VAP Prevention in ICU by BACTIGUARD coAting of endotracheaL Tube
Brief Title: VITAL - VAP Prevention by BIP (Bactiguard Infection Protection) ETT Evac in Belgian ICUs
Acronym: VITAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bactiguard AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PL-13674
Record Dates: First submitted 2020-01-13; First posted 2020-01-27 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Ventilator-associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Controlled study. Two interventions:
  1. Endotracheal tube with evacuation lumen without Bactiguard coating.
  2. Endotracheal tube with evacuation lumen with Bactiguard coating.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded, the two devices have the same appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Endotracheal tube with evacuation lumen without Bactiguard coating.
  Interventions: Device: ETTEvac
- Experimental group (Experimental): Endotracheal tube with evacuation lumen with Bactiguard coating.
  Interventions: Device: BIP ETTEvac

INTERVENTIONS:
Device: ETTEvac — Endotracheal tube with evacuation lumen without noble metal coating
  Arms: Control group
Device: BIP ETTEvac — Endotracheal tube with evacuation lumen with noble metal coating
  Arms: Experimental group

SUMMARY:
The study objective is to determine VAP (Ventilator Associated Pneumonia) baseline incidence in the ICU in patients receiving endotracheal tubes with evacuation lumen with and without Bactiguard coating. The study is randomized, prospective, controlled and blinded. All adult patients hospitalized in the ICUs from two tertiary hospitals (i.e.: Centre Hospitalier Universitaire Sart Tilman Liège , Centre Hospitalier Chrétien de Liège) and considered to be ventilated for more than 24 hours will be eligible to participate in the study.

DETAILED DESCRIPTION:
The aim of the study is to determine VAP (Ventilator Associated Pneumonia) baseline incidence in the ICU in patients receiving endotracheal tubes with evacuation lumen with and without Bactiguard Infection Protection (BIP) coating.

VAP is likely to occur in 10-20% of patients who are ventilated for at least 48 hours. These patients face a mortality risk estimated to be twice as high compared with similar ICU patients without VAP. Furthermore, VAP results in an average excess length of ICU stay with high hospital cost.

Bactiguard has developed an endotracheal tube coated with a thin layer of non-releasing metals (gold, silver and palladium) firmly attached to the surface. This Bactiguard coating is tissue friendly and aims to achieve an optimal combination of anti-infective properties to reduce biofilm formation, colonization and subsequent respiratory infection. Bactiguard coated urinary products have been on market since 1995 (initially in US, then also in Japan & Europe) and used in a large number of clinical studies and evaluations, showing reduction of urinary tract infections and also antibiotics use. A BIP ETT (without evacuation lumen) clinical safety and tolerability study was performed at Karolinska University Hospital during 20128. The study showed that BIP ETT is safe, well tolerable and performs well in clinical settings.

The present study of BIP ETT with evacuation lumen is randomized, prospective, controlled and blinded. All adult ICU patients hospitalized in the ICUs from two tertiary hospitals (i.e.: Centre Hospitalier Universitaire Sart Tilman Liège , Centre Hospitalier Chrétien de Liège) and considered to be ventilated for more than 24 hours will be eligible to participate in the study. 300 patients in total will be used to determine baselines levels (150 in each group).

The study tubes will be available not only in the ICUs but also in the emergency department, including the emergency vehicles, and in every hospital wards. The study tubes will not be available in the operating rooms except in the Post Anesthesia Care Units (PACU) and Recovery rooms.

ELIGIBILITY:
Inclusion Criteria:

* intubation with a study tube and a presumed duration of ventilation for more than 24h,
* age > 18 y,
* signed informed consent

Exclusion Criteria:

* tracheostomized patient
* life expectancy less than 48h,
* previous participation in the study
* pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
VAP incidence | Up to 28 days after inclusion
  Ventilator Associated Pneumonia incidence

SECONDARY OUTCOMES:
Nosocomial infections | Up to 28 days after inclusion
  Incidence of any kind of nosocomial infection
VAT incidence | Up to 28 days after inclusion
  Ventilator Associated Tracheabronchitis incidence
Antibiotics consumption | Up to 28 days after inclusion
Duration of ventilation | Up to 28 days after inclusion
  Days of intubation with study tube
Duration of ICU and hospital stay | Up to 28 days after inclusion
Mortality | Up to 60 days after inclusion
Tracheal bacterial colonization | Up to 28 days after inclusion
  Incidence of tracheal bacterial colonization reaching a CFU Count 10^6 CFU/ml
VAC and iVAC | Up to 28 days after inclusion
  Ventilator associated Condition and infectious iVAC

OTHER OUTCOMES:
Evaluation of microbial data | Up to 28 days of intubation after inclusion
  Amount and type of bacteria, resistance pattern
Evaluation of durability of the coating metals at the surface during use | Up to 28 days of intubation after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Misset, MD,Prof., Principal Investigator — CHU, Liege; Belgium
Locations (2):
- Belgium (2):
  - Centre Hospitalier Universitaire Sart Tilman Liège, Liège
  - Centre Hospitalier Chrétien de Liège and Centre Hospitalier Chrétien (CHC Clinique de l'Espérance), Liège

REFERENCES:
- [Derived] Damas P, Legrain C, Lambermont B, Dardenne N, Guntz J, Kisoka G, Demaret P, Rousseau AF, Jadot L, Piret S, Noirot D, Bertrand A, Donneau AF, Misset B. Prevention of ventilator-associated pneumonia by noble metal coating of endotracheal tubes: a multi-center, randomized, double-blind study. Ann Intensive Care. 2022 Jan 4;12(1):1. doi: 10.1186/s13613-021-00961-y. PMID 34981245